CLINICAL TRIAL: NCT05146141
Title: The Relationship Between Bent-arm Throw and Tennis Performance
Brief Title: Bent-arm Throw and Tennis Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Physiotherapist, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Bent-arm throw in tennis
Record Dates: First submitted 2021-10-20; First posted 2021-12-06 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Tennis Serve Performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants will have to perform a bent-arm throw program 5 minutes before each training session
  Interventions: Other: Bent-arm throw exercises
- Control group (Sham Comparator): No intervention. They will perform their usual warm-up.
  Interventions: Other: Bent-arm throw exercises

INTERVENTIONS:
Other: Bent-arm throw exercises — The participants will have to perform bent-arm throw exercises 5 minutes before each training session

SUMMARY:
The objective of this study is to explore the relaitonship betwenn bent-arm throw and tennis serve performance.

Young players (9-12 years) will be assessed at the beginning of the season and at mid-season to measure the accuracy, the speed and the gesture of tennis serve. During a mid-season, they will have to perform a bent-arm throw warm-up program 5 minutes before each training session to increase their ability to throw.

ELIGIBILITY:
Inclusion Criteria:

* age between 9 and 12
* playing tennis at least 2 times a week

Exclusion Criteria:

* history of shoulder injury or shoulder pain

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Serve velocity | change between the beginning and the end of the season (6 months)
  Serve velocity will be assessed with a radar
Serve precision | change between the beginning and the end of the season (6 months)
  Serve accuracy will be measured with a target placed on the field
Serve bidimensional movement | change between the beginning and the end of the season (6 months)
  serve gesture will be analysed with camera's

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No